CLINICAL TRIAL: NCT02890784
Title: Treatment Optimization for Patients With Chronic Myeloid Leukemia (CML) With Treatment naïve Disease (1st Line) and Patients With Resistance or Intolerance Against Alternative Abl-Kinase Inhibitors (≥2nd Line)
Brief Title: Dasatinib Holiday for Improved Tolerability
Acronym: DasaHIT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Jena (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Andreas Hochhaus, Director of the Clinic of Internal Medicine II, University of Jena
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DasaHIT
Record Dates: First submitted 2016-01-14; First posted 2016-09-07 (Estimated); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Myeloid Leukemia, Chronic
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A. Standard arm (Active Comparator): 100mg dasatinib (SPRYCEL®) daily dose (QD) (7x100) (Standard therapy)
  Interventions: Drug: dasatinib (SPRYCEL®)
- B. Study arm (Experimental): 100mg dasatinib (SPRYCEL®) (QD) weekdays (1-5) only (5x100+2x0) (overall dose reduction per week)
  Interventions: Drug: dasatinib (SPRYCEL®)

INTERVENTIONS:
Drug: dasatinib (SPRYCEL®) — Treatment optimization for patients with chronic myeloid leukemia (CML)

SUMMARY:
Treatment optimization for patients with chronic myeloid leukemia (CML) with treatment naïve disease (1st line) and patients with resistance or intolerance against alternative Abl-Kinase Inhibitors (≥2nd line) (DasaHIT Trial (Dasatinib Holiday for Improved Tolerability))

DETAILED DESCRIPTION:
Dasatinib is indicated in Europe for:

* Treatment of adult patients with newly diagnosed Philadelphia chromosome positive (Ph+) chronic myeloid leukemia (CML) in the chronic phase
* Chronic, accelerated or blast phase CML with resistance or intolerance to prior therapy including imatinib
* Ph+ acute lymphoblastic leukemia (ALL) and lymphoid blast CML with resistance or intolerance to prior therapy Compared to imatinib, dasatinib in CML achieves faster and better responses. Dasatinib is known for its selected toxicities (fluid retention, edema, pleural effusion, and hematological toxicity) requiring dose reductions or treatment interruptions; these toxicities are more frequent in the first two years of treatment. A randomized dose optimization trial for QD dosing vs. BID dosing has demonstrated non-inferiority with regards to efficacy with an improved toxicity profile. In a pilot study, analyzing patients with dasatinib toxicity, a fixed dasatinib weekend holiday allowed safe toxicity management without impairing efficacy. Furthermore the alternated schedule was also able to improve response parameters in patients that had never achieved an acceptable response prior to the onset of dasatinib holiday dosing schedule. The biological rationale for a holiday dosing schedule is that dasatinib has shown an improved cell death of CML cells even after short exposure times; this improved cell death exceeds the killing rate observed with imatinib in vitro. In summary, the reported preclinical and clinical evidence indicates that efficacy seems to require adequate dasatinib Cmax, while low Cmin (five half-lives between doses) does not impair efficacy nor induces drug resistance. It is speculated that a weekend holiday, allowing a better tolerability, would improve patients' drug adherence. The Investigators hypothesize that a dasatinib holiday schedule (5x100mg+2x0mg weekly) compared to a regular dose (7x100mg weekly) will reduce the rate of clinically significant toxicity (e.g., fluid retention, hematological toxicity, musculoskeletal pain) by 20% observed within the first two years of treatment. The Investigators also hypothesize that the dasatinib holiday schedule is non-inferior to dasatinib regular dose in achieving the European LeukemiaNet (ELN) recommended levels of response within the first 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with diagnosis of CP-CML with cytogenetic confirmation of Ph+ chromosome [t(9;22)(q34;q11)].
* Ph negative cases or patients with variant translocations who are BCR-ABL positive in multiplex PCR4 will be also considered eligible.
* ECOG performance status ≤2.
* Age ≥ 18 years old (no upper age limit is given)
* Serum levels of potassium, magnesium and total calcium within the normal limits (≥LLN [lower limit of normal] and ≤ULN [upper limit of normal]). Correction of electrolytes' levels with supplements to meet enrolment criteria is allowed.
* AST and ALT ≤2.5 x ULN or 5.0 x ULN if considered due to leukemia
* Alkaline phosphatase ≤2.5 x ULN unless considered due to leukemia
* Total bilirubin ≤1.5 x ULN, except known Gilbert disease
* Serum creatinine ≤2 x ULN
* Written informed consent prior to any study procedures being performed.

For 1st-line patients:

• Pre-treatment with hydroxyurea up to 6 months and imatinib or dasatinib for duration of up to 4 weeks is permitted.

For ≥ 2nd-line patients:

• Patients with treatment failure according to the 2013 ELN Recommendations criteria3 or treatment intolerance as assessed by the investigator after prior treatment with TKIs other than dasatinib (imatinib, nilotinib, bosutinib, ponatinib).

Exclusion Criteria:

* Previous allogeneic stem cell transplantation (AlloSCT)
* Known impaired cardiac function, including any of the following:

  * Congenital long QT syndrome
  * History of or presence of clinically significant ventricular or atrial tachyarrhythmia
  * QTc >450 msec on screening ECG
  * Myocardial infarction within 6 months prior to starting therapy
* Other clinical significant heart disease (e.g. unstable angina pectoris, congestive heart failure)
* Acute or chronic viral hepatitis with moderate or severe hepatic impairment (Child-Pugh scores >6), even if controlled
* Other concurrent uncontrolled medical conditions (e.g., active or uncontrolled infections, acute or chronic liver and renal disease) that could cause unacceptable safety risks or compromise compliance with the protocol
* Impaired gastrointestinal function or disease that may alter the absorption of study drug (e.g., ulcerative disease, uncontrolled nausea, vomiting and diarrhea, malabsorption syndrome, small bowel resection or gastric by-pass surgery)
* Concomitant medications known to be strong inducers or inhibitors of the CYP450 isoenzyme CYP3A4
* Patients who have undergone major surgery ≤2 weeks prior to starting study drug or who have not recovered from side effects of such therapy
* Patients who are pregnant or breastfeeding or women of reproductive potential not employing an effective method of birth control. Women of childbearing potential must have a negative serum pregnancy test within 14 days prior to administration of dasatinib. Post-menopausal women must be amenorrheic for at least 12 months in order to be considered of non-childbearing potential. Male and female patients must agree to employ an effective method of birth control throughout the study and for up to 3 months following discontinuation of study drug
* Known diagnosis of human immunodeficiency virus (HIV) infection (HIV testing is not mandatory)
* Active autoimmune disorder, including autoimmune hepatitis
* Known serious hypersensitivity reactions to dasatinib
* Patients with a history of another primary malignancy that is currently clinically significant or currently requires active intervention
* Patients unwilling or unable to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 291 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
cumulative toxicity score | month 24
  The cumulative toxicity score after two years of dasatinib treatment. More specifically, toxicity will be assessed taking into account both the rate of grade 2-4 toxicities and the cumulative severity of adverse events of specific interest. The following AEs of specific interest will be used to compose the cumulative toxicity score:
  1. Pleural effusion
  2. Fluid retention, other (edema, pericardial effusion, pulmonary arterial hypertension, congestive heart failure, pulmonary edema)
  3. Hematological toxicity (neutropenia, thrombocytopenia, anemia)
  4. Others (Musculoskeletal pain, skin toxicity (rash), gastrointestinal toxicity (nausea, diarrhea, abdominal pain, vomiting)
Rate of molecular Response | month 24
  The co-primary endpoint of the study is: rate of major molecular response (MMR) as assessed by BCR-ABL (IS [International Score] in %) -monitoring by 24 months to safeguard non-inferiority of the test cohort.

SECONDARY OUTCOMES:
Quality of life assessment | month 24
  Quality of life assessment via Patient-Questionnaire.
Rate of molecular Response | 6 and 12 months
  Rate of molecular response (MMR)as assessed by BCR-ABL (IS [International Score] in %) at 6 and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Hochhaus, Prof., Principal Investigator — Jena University Hospital
Locations (53):
- Germany (53):
  - Uniklinik der RWTH Aachen, Aachen
  - Gesundheitszentrum St. Marien GmbH, Amberg
  - Gemeinschaftspraxis Dres. Klausmann, Aschaffenburg
  - OnkoBer, Berlin
  - Evangelisches Klinikum Bethel gGmbH, Bielefeld
  - Universitätsklinikum Bonn, Bonn
  - Klinikum Bremen-Mitte gGmbH, Bremen
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Gemeinschaftspraxis Mohm/Prange-Krex, Dresden
  - Universitätsklinikum Carl Gustav Carus an der Technischen Universität Dresden, Dresden
  - Helios St. Johannes Klinik Duisburg, Duisburg
  - Gemeinschaftspraxis Erlangen, Erlangen
  - Universitätsklinikum Essen, Essen
  - Universitätsklinikum Frankfurt, Frankfurt
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Katholisches Karl-Leisner Klinikum, Goch
  - MVZ Onkologische Kooperation Harz, Goslar
  - ConMed GmbH, Göttingen
  - Hämato-Onkologische Gemeinschaftspraxis Halberstadt, Halberstadt
  - Universitätsklinikum Halle/S., Halle
  - Asklepios MVZ Onkologie, Hamburg
  - MediProjekt GbR, Hanover
  - St. Bernward Krankenhaus Hildesheim, Hildesheim
  - Universitätsklinikum Jena, Jena
  - Institut für med. Dokumentation, Gutachtenstellung, Gesundheitsförderung und Qualitätssicherung GbR, Kaiserslautern
  - Städtisches Klinikum Karlsruhe gGmbH, Karlsruhe
  - St. Vincentius-Kliniken Karlsruhe, Karlsruhe
  - Onkologische Gemeinschaftspraxis, Kassel
  - Klinikum Kassel, Kassel
  - Städtisches Krankenhaus Kiel GmbH, Kiel
  - Universitätsklinikum Schleswig-Holstein, Kiel
  - InVo Institut für Versorgungsforschung, Koblenz
  - MVZ Hämatologie und Onkologie, Krefeld
  - Onkologische Schwerpunktpraxis, Kronach
  - Onkologisches Zentrum, Lebach
  - Studienzentrum UnterEms, Leer
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsmedizin Mannheim, Mannheim
  - Universitätsklinikum Gießen und Marburg GmbH, Marburg
  - Stauferklinikum Schwäbisch Gmünd, Mutlangen
  - Rotkreuzklinikum München, München
  - Gemeinschaftspraxis Hämatologie/ Onkologie, München
  - Universitätsklinikum Münster, Münster
  - Hämatologisch-onkologische Schwerpunktpraxis, Neustadt am Rübenberge
  - Klinikum Passau, Passau
  - Kreiskliniken Reutlingen GmbH, Reutlingen
  - Universitätsmedizin Rostock, Rostock
  - Klinikum Südstadt Rostock, Rostock
  - Hämatologie-Onkologie Stolberg, Stolberg
  - Klinikum Mutterhaus der, Trier
  - Universitätsklinikum Ulm, Ulm
  - Schwarzwald-Baar Klinikum Villingen-Schwenningen GmbH, Villingen-Schwenningen
  - Rems-Murr-Klinik Winnenden, Winnenden

IPD SHARING:
Plan to Share IPD: No